CLINICAL TRIAL: NCT02989558
Title: A Prospective, Multicentre, Randomized, Open Label, Blinded Endpoint, Phase 3 Trial to Assess the Safety and Efficacy of Prophylactic TicagrelOr With Acetylsalicylic Acid Versus CLopidogrel With Acetylsalicylic Acid in the Development of Cerebrovascular EMbolic Events During Transcatheter Aortic Valve Implantation (TAVI) OperationS - the PTOLEMAIOS Study.
Brief Title: A Trial to Assess the Safety and Efficacy of Prophylactic TicagrelOr With Acetylsalicylic Acid Versus CLopidogrel With Acetylsalicylic Acid in the Development of Cerebrovascular EMbolic Events During TAVI
Acronym: PTOLEMAIOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Dr. Emmanouil Vavouranakis, Associate Professor, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D5130C00173
Record Dates: First submitted 2016-12-03; First posted 2016-12-12 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Ticagrelor; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ticagrelor plus ASA (Active Comparator): Subjects in the Ticagrelor group will receive ASA 80mg qd 7 days prior to the TAVI procedure and for 90 days and Ticagrelor 90mg bid 1 day prior to the TAVI procedure and for 90 days.
  Interventions: Drug: Ticagrelor plus ASA
- Clopidogrel plus ASA (Active Comparator): Subjects in the Clopidogrel group will receive ASA 80mg qd 7 days prior to the TAVI procedure and for 90 days and Clopidogrel as a loading dose of 300 mg 1 day prior to the TAVI procedure and thereafter 75mg qd for 90 days.
  Interventions: Drug: Clopidogrel plus ASA

INTERVENTIONS:
Drug: Ticagrelor plus ASA — Subjects in the Ticagrelor group will receive ASA 80mg qd 7 days prior to the TAVI procedure and for 90 days and Ticagrelor 90mg bid 1 day prior to the TAVI procedure and for 90 days.
  Other Names: Brilique plus aspirin
  Arms: Ticagrelor plus ASA
Drug: Clopidogrel plus ASA — Subjects in the Clopidogrel group will receive ASA 80mg qd 7 days prior to the TAVI procedure and for 90 days and Clopidogrel as a loading dose of 300 mg 1 day prior to the TAVI procedure and thereafter 75mg qd for 90 days.
  Other Names: Clopidogrel plus aspirin
  Arms: Clopidogrel plus ASA

SUMMARY:
Ticagrelor administered with Acetylsalicylic Acid (ASA) will provide better cerebral protection from microembolization in the cerebral circulation during Transcatheter Aortic Valve Implantation (TAVI) and 30 days afterwards, than Clopidogrel plus ASA. This hypothesis will be investigated by measuring the number of High Intensity Transient Signals (HITS) as assessed with transcranial Doppler (TCD) on middle cerebral arteries.

DETAILED DESCRIPTION:
TAVI has recently provided a therapeutic alternative to patients with symptomatic aortic stenosis who are inoperable or at high-risk for surgical valve replacement.

It has been documented with MRI studies that >70% of the patients undergoing TAVI develop new cerebral infarct lesions. Of these, only a ~3% to ~ 6% represent clinical significant events (transient ischemic attacks, disabling and non-disabling stroke). With the expected expansion of TAVI in lower risk patients and younger age even silent cerebral lesions will be of major importance [7], thus ways to overcome or decrease it will have a rapid and wide penetration.

Clinically apparent or "silent" stroke during TAVI may be attributed to a range of different mechanisms. The source of a cerebral ischemia during TAVI is multifactorial. One of the proposed mechanisms is the increased risk of thrombus formation both on the aortic atherosclerotic plaques and on bioprosthetic valve frame and tissue due to inadequate platelet inhibition during or after TAVI. Furthermore, high residual platelet reactivity in the presence of incomplete endothelial coverage of the valve following TAVI may promote formation of fibrin/platelet thrombi. Other mechanisms involve embolization from a variety of origins i.e. atheroembolism from the ascending aorta or aortic arch, calcific emboli from the aortic valve, thromboembolism from catheters.

Platelets are the main target of preventative therapy against cerebral ischemic events, owing to the observation that, in addition to promoting arterial thrombosis, platelets have a key role in various nonthrombotic, inflammatory pathways of plaque progression The clinical apparent or "silent" embolic events may be recognized with TCD performed during TAVI as documented in published clinical studies. TCD is an accepted surveillance technique during neurological interventions (such as TAVI, atrial septal defects/patent form ovale closure, carotid endarterectomy). Moreover, studies utilizing TCD during TAVI for evaluation of potential embolization are available. TCD observes HITS that may be quantified and potentially correlated with neurological events. However, it should be noted that this approach is not able to discriminate the exact source or composition of the emboli The use of embolic protection devices (e.g. the Embrella Embolic Deflector system) during TAVI surprisingly showed an increase in the number of cerebral ischemic lesions on postprocedural brain imaging when compared to dual antiplatelet therapy.

The first few days post TAVI carry the highest risk for a thromboembolic event, thus special therapeutic and diagnostic approaches should be taken into consideration when regarding this procedure. Similarly, surgical bioprosthetic valve implantation has shown to have a higher risk of thromboembolic events within 3 months of the procedure.

The administration of a monotherapy with ASA after biological aortic valve replacement failed to show improvement in the incidence of thromboembolic events. Dual antiplatelet therapy is traditionally started prior to TAVI and continued for 6 months. Nevertheless, in these fragile elderly patients dual antiplatelet therapy increases the risk of haemorrhage. In addition the protection achieved by these agents is questionable and resistance to aspirin and Clopidogrel has been observed in a high percentage.

Platelet Function Testing has been proven to characterize the patients at high risk for adverse outcome after percutaneous coronary interventions. However, pharmacological interventions to overcome this increased risk have not been established.

The use of Ticagrelor has been proven to reduced cerebral ischemic events in acute coronary syndromes (ACS) without significantly increasing the major bleeding complications, despite the more potent antithrombotic effect. Moreover, total mortality was substantially decreased using Ticagrelor, as the risk of intracranial hemorrhage or fatal stroke was low.

In the DISPERSE-2 Trial, slightly higher rates of minor bleeding where observed with Ticagrelor compared to Clopidogrel; however major bleeding events were lower with Ticagrelor. Overall, total bleeding events were similar in the Ticagrelor and Clopidogrel groups, as well as in patients with additional antithrombotic agents or undergoing invasive procedures. However, the administration of Ticagrelor allows for greater flexibility and safety if the need for discontinuation of antiplatelet agents should arise, as it has a half life of only 12 hours [16]. More importantly, Ticagrelor is a reversible platelet inhibitor, in contrast to Clopidogrel and ASA who bind irreversibly to platelet cell membrane receptors and the cyclooxygenase enzyme respectively, and whose effects persist for duration of the platelet life span. Therefore, in case of a bleeding event where antiplatelet therapy needs to be deescalated, monotherapy with Ticagrelor could prove to be the safer option.

Ticagrelor has been documented to demonstrate faster onset and more potent inhibition of platelet aggregation than Clopidogrel. These properties of Ticagrelor may contribute to lower rates of thrombotic outcomes compared to Clopidogrel. However, bleeding events are a concern with the more potent antiplatelet agents Ticagrelor and Prasugrel. This risk of bleeding is correlated to the concomitant dosage of ASA, therefore the lowest effective dose of 80mg of ASA was chosen as a background therapy for this study.

Compared to Prasugrel, another thienopyridine drug, Ticagrelor has shown to provide a more potent effect on the microcirculation of patients undergoing percutaneous coronary intervention.

Moreover, the use of current antiplatelet regimens during and post TAVI has not been well established by clinical data. Currently, there are no guidelines regarding antiplatelet pre- treatment before TAVI. The European Society of Cardiology practice guidelines (2012) suggest that in real-life double antiplatelet regimens are prescribed in the early post-TAVI period, without further issuing a specific recommendation. Even as such and with the wide clinical use of dual antiplatelet therapy perioperatively for TAVI, cases of thrombus formation on bioprosthetic valves have been documented. The manufacturer has attributed these events to suboptimal operative placement of the bioprosthesis, therefore caution must be taken in the positioning of the bioprosthetic valves in order to reduce the formation of emboli that could potentially cause a clinically significant cerebral ischemic event. The use of a more potent dual antiplatelet regimen with Ticagrelor could prove more efficient in this aspect.

The present study aims to evaluate whether platelet inhibition with one new antiplatelet agent provides better cerebral protection from microembolization in the cerebral circulation during TAVI, than the currently used Clopidogrel. We hypothesize that treatment with Ticagrelor plus ASA vs. Clopidogrel plus ASA in patients undergoing TAVI will result in fewer HITS as assessed with TCD on middle cerebral arteries.

This is the first study to directly compare treatment with Ticagrelor with Acetylsalicylic vs. Clopidogrel with Acetylsalicylic regimen in subjects undergoing TAVI regarding cerebral embolic events as assessed with TCD of both middle cerebral arteries. If significant reduction in HITS number in the Ticagrelor group is proven, this will implicate a possible way to decrease in cerebral ischemic lesions in TAVI subjects. Undoubtedly, as TAVI candidates are increasing in number and decreasing in age, the prevention of neurological consequences is of paramount importance.

ELIGIBILITY:
Inclusion Criteria:

1. The subject (or where unable to do so, their legally acceptable representative) must be able to provide written informed consent prior to any study specific criteria, stating that he or she understands the purpose of and the procedures required for the study and is willing to participate in the study.
2. Female and/or male subjects aged 18 years or older.
3. High risk (EuroSCOREa ≥18, or considered inoperable) for surgical aortic valve replacement.
4. Is expected to benefit from the placement of TAVI.
5. Does not suffer from any disease or condition that would limit his/her life expectancy of <6 months.
6. The subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.
7. Subjects must meet the following laboratory results from Visit 0 for study inclusion:

   1. Hemoglobin ≥ 10 g/dL
   2. Platelets ≥ 100 X 103 cells/μL
   3. Absolute neutrophil count (ANC) ≥ 1000 cells/μL
   4. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) levels must be within 1.5 times the upper limit of normal (ULN) range for the laboratory conducting the test.
   5. Total bilirubin ≤ 2x ULN.

Exclusion Criteria:

1. Have scheduled any elective surgery in the next 4 months following screening procedures.
2. History of hypocoagulopathy.
3. Previous thromboembolism or known hypercoagulopathy (acquired or congenital).
4. Antiplatelet therapy, other than ASA, within 7 days before randomization that cannot be discontinued due to the underlying disease.
5. History of gastric or duodenal ulcer disease verified by endoscopy or barium meal double-contrast technique within the 3 months.
6. Moderate or severe hepatic impairment.
7. Known hypersensitivity to any of the investigational products or their components.
8. Presence of any other clinically significant disease or disorder which, in the opinion of the Investigator (by its nature or by being inadequately controlled), might put the subject at risk due to participation in the study, or may influence the conduct or the interpretation of the results of the study or the subject's ability to complete the study.
9. Any identified contraindication for using Ticagrelor, Clopidogrel or ASA.
10. History or recent findings of atrial fibrillation.
11. Significant carotid artery disease on either internal carotid artery, as defined by a >50 % diameter reduction on carotid ultrasonography.
12. Unwillingness to receive or intolerant to any blood products.
13. Previous trauma or surgery to either femoral vein.
14. Major surgical procedure or trauma within the 30 days prior to enrolment.
15. Mechanical heart valve (any location).
16. Mitral or aortic bioprosthetic valve.
17. The subject is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator.
18. Reproductive status:

    1. Women who are pregnant or planning a pregnancy within 1 month of the end of study;
    2. Women who are breastfeeding;
    3. Women of childbearing potential who are unwilling or unable to use two highly effective methods of birth control to avoid pregnancy for the entire study period, as evaluated by the Investigator. Women who are not of childbearing potential are those that have a history of hysterectomy, bilateral oophorectomy, or are postmenopausal with no history of menstrual flow for ≥ 12 months prior to the screening Visit.

    Highly effective methods of birth control are defined as:

    Hormonal: established use of oral, implantable, injectable, or transdermal hormonal methods of conception; Placement of an intrauterine device; Placement of an intrauterine system; Mechanical/barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) in conjunction with spermicide (foam, gel, film, cream or suppository); When used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides provides more effective birth control. However, spermicides alone may not be effective in preventing pregnancy and must be used with a barrier such as a condom or diaphragm.

    Surgical sterilization of male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate; for female patients on the study, the vasectomized male partner should be the sole partner for that patient) in conjunction with spermicide, condom, or diaphragm; Sexual true abstinence: when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
19. International normalized ratio (INR) ≥ 2 on the day before the TAVI procedure.
20. History of hemorrhagic stroke, intracranial, intraocular, spinal, retroperitoneal or atraumatic intra-articular hemorrhage, intracerebral mass or aneurysm, or arteriovenous malformation.
21. Severe left ventricular dysfunction (left ventricular ejection fraction<15%).
22. Severe aortic regurgitation or mitral regurgitation, according to the 2012 European Society of Cardiology and the European Association for Cardio-Thoracic Surgery guidelines (See Appendix 16)
23. Hemodynamic instability (e.g. requiring inotropic or intra-aortic balloon pump support) within 2 hours of the procedure.
24. Subject is dialysis dependent.
25. Any condition requiring the use of anticoagulants that cannot be stopped for the duration of the study.
26. Acute myocardial infarction, major surgery or any therapeutic cardiac procedure (other than balloon aortic valvuloplasty) within 30 days.
27. Gastrointestinal or genitourinary bleed within 30 days.
28. Absolute contraindications or allergy to iodinated contrast that cannot be pre-medicated.
29. Treatment with other investigational drugs (including investigational vaccines) or devices within the 30 days preceding enrolment or planned use of other investigational drugs or devices before the end of the study.
30. Known alcohol or drug abuser.
31. The subject has received any prohibited therapies, as defined in Section 5.7 before the planned first dose of investigational product or is scheduled to receive during the study period. These include, but are not limited to: strong cytochrome P450 3A (CYP3A) inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, erythromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, over 1 litre daily of grapefruit juice), CYP3A substrates with a narrow therapeutic index (cyclosporine, quinidine, simvastatin at doses >40 mg daily, lovastatin at doses >40 mg daily), and strong CYP3A inducers (rifampin/rifampicin, phenytoin, carbamazepine, phenobarbital).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
The number of confirmed HITS, as assessed by Transcranial Doppler (TCD), between the two treatment groups during the TAVI procedure. | During the TAVI procedure
  The primary objective is to identify any potential differences between the two treatment groups, subjects receiving Ticagrelor with ASA vs. those receiving Clopidogrel with ASA, in preventing cerebrovascular embolic events during the TAVI procedure, as assessed by measuring the number of HITS with an operative transcranial continuous-function Doppler.

SECONDARY OUTCOMES:
The incidence of cerebral embolic events between the two treatment groups, as assessed by HITS measured by TCD at subject discharge. | At day 5, an average at discharge. Data about HITS
  The differences in the incidence of cerebral embolic events between the two treatment groups, as assessed by HITS measured by TCD at subject discharge.
the incidence of cerebral embolic events in each treatment group, during the TAVI procedure, and at subject discharge. | At day 1, procedure day and at day 5, an average at discharge. Data about HITS
  The differences in the incidence of cerebral embolic events in each treatment group, as assessed by HITS measured by TCD preoperatively, during the TAVI procedure, and at subject discharge.
The differences between the two treatment groups in induced platelet inhibition, at the day of the procedure. | At day 1, procedure day. Data about platelet inhibition
  The differences between the two treatment groups in induced platelet inhibition, as assessed by the use of the P2Y12 VerifyNow® assay at the day of the procedure.
The differences between the two treatment groups in induced platelet inhibition, at subject discharge. | At day 5, an average at discharge. Data about platelet inhibition
  The differences between the two treatment groups in induced platelet inhibition, as assessed by the use of the P2Y12 VerifyNow® assay at subject discharge.

CONTACTS AND LOCATIONS:
Overall Officials: EMMANOUIL VAVOURANAKIS, Ass. Prof, Principal Investigator — University of Athens, 1st Department of Cardiology, Hippokration Hospital
Locations (1):
- 1st Department of Cardiology, Hippokration Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Storey RF, Husted S, Harrington RA, Heptinstall S, Wilcox RG, Peters G, Wickens M, Emanuelsson H, Gurbel P, Grande P, Cannon CP. Inhibition of platelet aggregation by AZD6140, a reversible oral P2Y12 receptor antagonist, compared with clopidogrel in patients with acute coronary syndromes. J Am Coll Cardiol. 2007 Nov 6;50(19):1852-6. doi: 10.1016/j.jacc.2007.07.058. Epub 2007 Oct 23. PMID 17980251
- [Background] Kowalczyk M, Banach M, Mikhailidis DP, Hannam S, Rysz J. Ticagrelor--a new platelet aggregation inhibitor in patients with acute coronary syndromes. An improvement of other inhibitors? Med Sci Monit. 2009 Dec;15(12):MS24-30. PMID 19946242
- [Background] Husted S, Emanuelsson H, Heptinstall S, Sandset PM, Wickens M, Peters G. Pharmacodynamics, pharmacokinetics, and safety of the oral reversible P2Y12 antagonist AZD6140 with aspirin in patients with atherosclerosis: a double-blind comparison to clopidogrel with aspirin. Eur Heart J. 2006 May;27(9):1038-47. doi: 10.1093/eurheartj/ehi754. Epub 2006 Feb 13. PMID 16476694
- [Background] Dobesh PP, Oestreich JH. Ticagrelor: pharmacokinetics, pharmacodynamics, clinical efficacy, and safety. Pharmacotherapy. 2014 Oct;34(10):1077-90. doi: 10.1002/phar.1477. Epub 2014 Aug 28. PMID 25164528
- [Background] Ghanem A, Muller A, Nahle CP, Kocurek J, Werner N, Hammerstingl C, Schild HH, Schwab JO, Mellert F, Fimmers R, Nickenig G, Thomas D. Risk and fate of cerebral embolism after transfemoral aortic valve implantation: a prospective pilot study with diffusion-weighted magnetic resonance imaging. J Am Coll Cardiol. 2010 Apr 6;55(14):1427-32. doi: 10.1016/j.jacc.2009.12.026. Epub 2010 Feb 24. PMID 20188503
- [Background] Samim M, Agostoni P, Hendrikse J, Budde RP, Nijhoff F, Kluin J, Ramjankhan F, Doevendans PA, Stella PR. Embrella embolic deflection device for cerebral protection during transcatheter aortic valve replacement. J Thorac Cardiovasc Surg. 2015 Mar;149(3):799-805.e1-2. doi: 10.1016/j.jtcvs.2014.05.097. Epub 2014 Oct 17. PMID 25455466
- [Background] Rodes-Cabau J, Kahlert P, Neumann FJ, Schymik G, Webb JG, Amarenco P, Brott T, Garami Z, Gerosa G, Lefevre T, Plicht B, Pocock SJ, Schlamann M, Thomas M, Diamond B, Merioua I, Beyersdorf F, Vahanian A. Feasibility and exploratory efficacy evaluation of the Embrella Embolic Deflector system for the prevention of cerebral emboli in patients undergoing transcatheter aortic valve replacement: the PROTAVI-C pilot study. JACC Cardiovasc Interv. 2014 Oct;7(10):1146-55. doi: 10.1016/j.jcin.2014.04.019. PMID 25341709
- [Background] Brueck M, Kramer W, Vogt P, Steinert N, Roth P, Gorlach G, Schonburg M, Heidt MC. Antiplatelet therapy early after bioprosthetic aortic valve replacement is unnecessary in patients without thromboembolic risk factors. Eur J Cardiothorac Surg. 2007 Jul;32(1):108-12. doi: 10.1016/j.ejcts.2007.03.031. Epub 2007 Apr 20. PMID 17449264
- [Background] Cannon CP, Husted S, Harrington RA, Scirica BM, Emanuelsson H, Peters G, Storey RF; DISPERSE-2 Investigators. Safety, tolerability, and initial efficacy of AZD6140, the first reversible oral adenosine diphosphate receptor antagonist, compared with clopidogrel, in patients with non-ST-segment elevation acute coronary syndrome: primary results of the DISPERSE-2 trial. J Am Coll Cardiol. 2007 Nov 6;50(19):1844-51. doi: 10.1016/j.jacc.2007.07.053. Epub 2007 Oct 23. PMID 17980250
- [Background] Topol EJ, Easton D, Harrington RA, Amarenco P, Califf RM, Graffagnino C, Davis S, Diener HC, Ferguson J, Fitzgerald D, Granett J, Shuaib A, Koudstaal PJ, Theroux P, Van de Werf F, Sigmon K, Pieper K, Vallee M, Willerson JT; Blockade of the Glycoprotein IIb/IIIa Receptor to Avoid Vascular Occlusion Trial Investigators. Randomized, double-blind, placebo-controlled, international trial of the oral IIb/IIIa antagonist lotrafiban in coronary and cerebrovascular disease. Circulation. 2003 Jul 29;108(4):399-406. doi: 10.1161/01.CIR.0000084501.48570.F6. Epub 2003 Jul 21. PMID 12874182
- [Background] Alexopoulos D, Moulias A, Koutsogiannis N, Xanthopoulou I, Kakkavas A, Mavronasiou E, Davlouros P, Hahalis G. Differential effect of ticagrelor versus prasugrel on coronary blood flow velocity in patients with non-ST-elevation acute coronary syndrome undergoing percutaneous coronary intervention: an exploratory study. Circ Cardiovasc Interv. 2013 Jun;6(3):277-83. doi: 10.1161/CIRCINTERVENTIONS.113.000293. Epub 2013 Jun 4. PMID 23735473
- [Background] Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Lung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M; ESC Committee for Practice Guidelines (CPG); Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC); European Association for Cardio-Thoracic Surgery (EACTS). Guidelines on the management of valvular heart disease (version 2012): the Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Eur J Cardiothorac Surg. 2012 Oct;42(4):S1-44. doi: 10.1093/ejcts/ezs455. Epub 2012 Aug 25. No abstract available. PMID 22922698
- [Background] Gurbel PA, Bliden KP, Hiatt BL, O'Connor CM. Clopidogrel for coronary stenting: response variability, drug resistance, and the effect of pretreatment platelet reactivity. Circulation. 2003 Jun 17;107(23):2908-13. doi: 10.1161/01.CIR.0000072771.11429.83. Epub 2003 Jun 9. PMID 12796140
- [Background] Butler K, Maya J, Teng R. Effect of ticagrelor on pulmonary function in healthy elderly volunteers and asthma or chronic obstructive pulmonary disease patients. Curr Med Res Opin. 2013 May;29(5):569-77. doi: 10.1185/03007995.2013.781502. Epub 2013 Apr 2. PMID 23448616
- [Background] Zafar MU, Farkouh ME, Fuster V, Chesebro JH. Crushed clopidogrel administered via nasogastric tube has faster and greater absorption than oral whole tablets. J Interv Cardiol. 2009 Aug;22(4):385-9. doi: 10.1111/j.1540-8183.2009.00475.x. Epub 2009 May 28. PMID 19496900
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Guyton RA, O'Gara PT, Ruiz CE, Skubas NJ, Sorajja P, Sundt TM 3rd, Thomas JD; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC guideline for the management of patients with valvular heart disease: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jun 10;63(22):2438-88. doi: 10.1016/j.jacc.2014.02.537. Epub 2014 Mar 3. No abstract available. PMID 24603192
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB; Valve Academic Research Consortium-2. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document. J Thorac Cardiovasc Surg. 2013 Jan;145(1):6-23. doi: 10.1016/j.jtcvs.2012.09.002. Epub 2012 Oct 16. PMID 23084102
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Erdoes G, Basciani R, Huber C, Stortecky S, Wenaweser P, Windecker S, Carrel T, Eberle B. Transcranial Doppler-detected cerebral embolic load during transcatheter aortic valve implantation. Eur J Cardiothorac Surg. 2012 Apr;41(4):778-83; discussion 783-4. doi: 10.1093/ejcts/ezr068. Epub 2011 Dec 1. PMID 22423058